CLINICAL TRIAL: NCT04412499
Title: Study of the Link Between Psychosocial Treatments and the Need of Pharmacological Treatments in Children With Attention Deficit Hyperactivity Disorder : a Retrospective Online Study for Parents
Brief Title: Study of the Link Between Psychosocial Treatments and the Need of Pharmacological Treatments in Children With Attention Deficit Hyperactivity Disorder
Acronym: OPTIME-TDAH
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0275
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Youths
Keywords: ADHD; treatment with methylphenidate; behavioral parent training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylphenidate + parent-training programm: Methylphenidate and participation in a parent-training programme
- Methylphenidate alone: Methylphenidate alone

SUMMARY:
The Attention Deficit and Hyperactivity Disorder (ADHD) is a frequent disorder in children and adolescents. The diagnosis is clinical with the input of several informants (child, family, teachers, …). ADHD is a risk factor for academic difficulties, school dropout, social isolation, injury, oppositional behaviour. In school-age children and adolescents having moderate to high or persistent impairment despite psycho-educational support and environmental modification, the first-line treatment is methylphenidate. Group or individual cognitive behavioural therapy for parents and/or children and adolescents is recommended for co-occurring disorders and persistent impairment. In France, the initiation of methylphenidate requires an annual hospital prescription by a paediatrician or psychiatrist, and a regular medical supervision (weight, heart rate, blood pressure, …). At least once a year, the indication of methyphenidate needs to be re-evaluated and confirmed at the hospital. In case of lack of efficiency and/or poor tolerance, therapeutic alternatives including non-psychostimulants should be considered.

A randomized controlled trial evaluated the dose of methylphenidate received over a period of 13 months. It was observed that the "combined treatment" group (methylphenidate + psychosocial treatments) received a lower average dose of methylphenidate than the "methylphenidate alone" group. These results are difficult to extrapolate to the general population, due to the study protocol (regular monitoring of ADHD symptoms with the aim of total remission).

For a global consideration of children's needs, it is important to better understand the interactions between these two therapeutic approaches.

To participate in the study, parents will have to complete an online questionnaire. This questionnaire contains anamnestic data collection, questionnaires to assess ADHD symptoms and parenting practices.

ELIGIBILITY:
Inclusion criteria:

- Children 6-18 years of age, diagnosed with ADHD, treated with methylphenidate for at least 6 months. Parents' online response between may and june 2020.

Exclusion criteria:

- Exclusion of respondants not caring for the child , refusal to participate

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with ADHD, treated by methylphenidate, from primary care and community sample.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Daily dose of methylphenidate (mg/kg) depending on participation in a parent-training programme | 1 day
  Daily dose of methylphenidate (mg/kg) depending on participation in a parent-training programme

CONTACTS AND LOCATIONS:
Overall Officials: Chrys Amiel, MD, PharmD, MSc, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC